CLINICAL TRIAL: NCT07354022
Title: A Multicenter, Open-label, Randomized Controlled Phase III Clinical Study Evaluating the Efficacy and Safety of HRS-8080 Combined With Dalpiciclib Versus Fulvestrant Combined With Dalpiciclib in Patients With Locally Advanced or Metastatic Breast Cancer Resistant to Adjuvant Endocrine Therapy.
Brief Title: A Study to Evluate Efficacy and Safety of HRS-8080 Combined With Dalpiciclib in Patients With Advanced or Metastatic Breast Cancer Resistant to Adjuvant Endocrine Therapy.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-301
Record Dates: First submitted 2026-01-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-8080 combined with Dalpiciclib (Experimental)
  Interventions: Drug: HRS-8080 Tablet ; Dalpiciclib Isethionate
- Fulvestrant combined with Dalpiciclib (Active Comparator)
  Interventions: Drug: Fulvestrant injection ;Dalpiciclib Isethionate

INTERVENTIONS:
Drug: HRS-8080 Tablet ; Dalpiciclib Isethionate — * HRS-8080 Tablet
  * Dalpiciclib Isethionate
  Arms: HRS-8080 combined with Dalpiciclib
Drug: Fulvestrant injection ;Dalpiciclib Isethionate — * Fulvestrant injection
  * Dalpiciclib Isethionate
  Arms: Fulvestrant combined with Dalpiciclib

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS-8080 combined with dalpiciclib versus fulvestrant combined with dalpiciclib in patients with locally advanced/metastatic breast cancer who had developed drug resistance to prior adjuvant endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 - 75 years old;
2. Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 to 1;
3. Patients with histologically confirmed locally advanced or metastatic breast cancer;
4. Patients with prior adjuvant endocrine resistance following curative-intent surgery;
5. Menstrual status: postmenopausal, perimenopausal, or premenopausal;
6. Presence of evaluable lesions;
7. Organ function must meet required criteria.

Exclusion Criteria:

1. Patients with rapidly progressing disease, as judged by the investigator to be unsuitable for endocrine therapy;
2. Patients who have previously received fulvestrant or other novel SERMs (excluding tamoxifen and toremifene);
3. Patients with uncontrolled brain metastases, carcinomatous meningitis, or spinal cord compression;
4. Patients with a history of clinically significant cardiovascular disease;
5. Participants who have not recovered from adverse effects caused by prior therapies;
6. Participants with a history of another malignancy within the past 5 years or currently having another malignancy;
7. Known hypersensitivity to HRS-8080, fulvestrant, dalpiciclib, or any of their components, etc.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Investigator assessed Progression free survival (PFS) | Up to 5 years.
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), or death from any cause during the study.

SECONDARY OUTCOMES:
Progression free survival (PFS) evaluated by the blinded independent central review (BICR) | Up to 5 years
Overall response rate (ORR) | Up to 5 years
Clinical benefit rate (CBR) | Up to 5 years
Duration of response (DOR) | Up to 5 years
Overall survival (OS) | Up to 8 years
The incidence and severity of adverse events (AEs) | Up to 5 years
The incidence and severity of serious adverse events (SAEs) | Up to 5 years
Number of participants with vital sign abnormalities over the course of the study. Vital signs include respiratory rate, pulse rate, systolic and diastolic blood pressure, and temperature | Up to 5 years
Number of participants with clinical laboratory test abnormalities for haematology and biochemistry parameters over the course of the study | Up to 5 years
Heart rate (beats per minute) measured by 12-lead electrocardiography. | Up to 5 years
QT interval (ms) measured by 12-lead electrocardiography. | Up to 5 years
  Eastern Cooperative Oncology Group (ECOG) performance status. ECOG performance status was measured on a 6 point grade scale.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
Plasma concentrations of HRS-8080 and dalpiciclib isethionate | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital Fifth Medical Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided